CLINICAL TRIAL: NCT05853965
Title: Combination Treatment of Belantamab Mafodotin and Venetoclax in Treatment of Relapsed and Refractory T(11;14) Multiple Myeloma (Phase I/IIa) the BELI(E)VE-Trial
Brief Title: Combination Treatment of Belantamab Mafodotin and Venetoclax in Treatment of Relapsed and Refractory T(11;14) Multiple Myeloma
Acronym: BELI(E)VE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BELI(E)VE Trial; 2021-001413-37 (EudraCT Number)
Record Dates: First submitted 2023-04-22; First posted 2023-05-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse
Keywords: t(11;14); venetoclax; belantamab mafodotin; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; venetoclax

STUDY DESIGN:
Intervention Model Description: Phase I: 3+3 Fibonacci design Phase II: single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Experimental): Belantamab Mafodotin 1.9 mg/kg Q6W Venetoclax 400mg QD
  Interventions: Drug: Belantamab mafodotin, Venetoclax
- Cohort 2 (Experimental): Belantamab Mafodotin 1.9 mg/kg Q6W Venetoclax 800mg QD
  Interventions: Drug: Belantamab mafodotin, Venetoclax
- Cohort 3 (Experimental): Belantamab Mafodotin 1.9 mg/kg Q6W Venetoclax 400mg QD Dexamethasone 40mg Q1W (20mg for subjects ≥ 75 years)
  Interventions: Drug: Belantamab mafodotin, Venetoclax
- Cohort 4 (Experimental): Belantamab Mafodotin 1.9 mg/kg Q6W Venetoclax 800mg QD Dexamethasone 40mg Q1W (20mg for subjects ≥ 75 years)
  Interventions: Drug: Belantamab mafodotin, Venetoclax

INTERVENTIONS:
Drug: Belantamab mafodotin, Venetoclax — Belantamab mafodotin (IV) Venetoclax (PO)

SUMMARY:
The goal of this clinical trial is to learn about the safety and efficacy of the drug combination belantamab mafodotin and venetoclax, with or without the addition of dexamethasone, in patients with relapsed/refractory multiple myeloma bearing the translocation t(11;14)

ELIGIBILITY:
Relapsed and refractory t(11;14) Multiple Myeloma (RRMM)

Inclusion criteria:

1. Subjects must be ≥ 18 years of age.
2. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
3. Subjects must voluntarily sign and date an in-formed consent form
4. Subjects must have had documented multiple myeloma requiring treatment as defined by the criteria below:

   Monoclonal plasma cells in the bone marrow > 10% and/or presence of a biopsy proven plasmacytoma at some point in their disease history requiring treatment according diag-nostic criteria (IMWG updated criteria 2014, Rajkumar et al. 2014) with measurable dis-ease at screening (serum M-protein > 500 mg/dL or urine M protein 200 mg/24h, in case of oligosecretory MM serum free light chain > 10mg/dL and abnormal kap-pa/lambda free light chain ratio)
5. Cytogenetics/FISH confirming t(11;14)
6. Prior treatment requirements:

   Prior treatment requirements:

   a. Subjects must have received at least 1 prior treatment line (induction, high-dose, consolidation and maintenance is considered as one treatment line). All patients have to have received at least one proteasome inhibitor and at least one immunomodulatory agent and at least one anti-CD38 monoclonal antibody.

   b. Subjects must have documented evidence of progressive disease on or after the last treatment line.

   c. Subjects with a history of autologous SCT are eligible for study participation provided the following eligibility criteria are met: i. ASCT was >100 days prior to initiating study treatment, and ii. No active bacterial, viral, or fungal in-fection(s) present.
7. Subjects must have adequate organ function, defined as follows:

   a. Hemoglobin ≥8.0 g/dL (without transfusion of red blood cells for the past 14 days) b. Absolute neutrophil count ≥ 1.5 x109/L (with-out growth factor support for the past 14 days) c. Platelet count more or equal 75 x109/L (with-out growth factor or platelet stimulating agents for the past 14 days) d. Adequate hepatic function per local laborato-ry reference range as follows: i. Aspartate aminotransferase (AST) ≤ 2,5 x upper limit of normal (ULN); ii. Alanine aminotransferase (ALT) ≤ 2.5 x ULN iii. Total bilirubin ≤ 1.5 x ULN, except in subjects with congenital bilirubinemia, such as Gilbert syndrome (direct bili-rubin ≤ 1.5 x ULN). Isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%.

   e. Subjects must have adequate renal function as demonstrated by eGFR ≥30 mL/min/ 1.73 m2 as calculated by Modified Diet in Renal Disease (MDRD) formula f. Spot urine (albumin/creatinine ratios (spot urine) <500 mg/g (56 mg/mmol) OR Urine Dipstick Negative/trace (if 1+ only eligible if confirmed <500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void) g. Corrected serum calcium ≤ 14 mg/dL (≤3,5 mmol/L); or free ionized calcium ˂ 6,5 mg/dL (˂1,6 mmol/L)
8. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

   1. Is not a woman of childbearing potential (WOCBP) OR
   2. Is a WOCBP and using a contraceptive method that is highly effective
9. Male participants are eligible to participate if they agree to the refrain from donating sperm and either bei abstinent from heterosexual intercourse or agree to use a highly effective contraceptive method during the intervention period and for 6 months after the last dose of study treatment to allow for clearance of any altered sperm
10. All subjects must agree to refrain from donating blood while on study drug and for 28 days after discontinuation from this study treatment.
11. All subjects must agree not to share study medication.
12. All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0) must be ≤ Grade 1 at the time of en-rolment except for alopecia.

Exclusion Criteria:

1. Subject has received prior Venetoclax and/or anti BCMA treatment.
2. Participant has used an investigational drug or approved systemic anti-myeloma therapy with-in 14 days or five half-lives, whichever is short-er, preceding the first dose of study drug. The only exception is emergency use of a short course of corticosteroids (equivalent of Dexa-methasone 40 mg/day for a maximum of 4 days) up to 7 days before treatment.
3. Participant has had plasmapheresis or radia-tion therapy within 7 days prior to first dose of study treatment
4. Participant has current corneal epithelial dis-ease except mild changes in corneal epitheli-um
5. Participant has current unstable liver or biliary disease
6. Participant has a presence of active renal con-dition (infection, requirement for dialysis or any other condition that could affect participant's safety).
7. Participant has had major surgery ≤ 4 weeks prior to initiating study treatment. Kyphoplasty is not considered a major surgery.
8. Participant must not use contact lenses while participating in this study. Bandage contacts may be prescribed by an eye care professional if needed.
9. Participant has any evidence of active mucosal or internal bleeding or other gastrointestinal disease that may significantly alter the absorp-tion of oral drugs.
10. Participant has evidence of cardiovascular risk as defined in the protocol
11. Participant has known immediate or delayed hypersensitivity reaction or idiosyncratic reac-tions to IMPs or drugs chemically related to IMPs, or any of the components of the study treatment
12. Participant has an invasive malignancy other than disease under study within 5 years before trial inclusion, except

    * Adequately treated in situ carcinoma of the cervix uteri or the breast;
    * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
    * Prostate cancer Gleason grade 6 or lower AND with stable Prostate Specific Antigen (PSA) levels off treatment;
    * Previous malignancy with no current evi-dence of disease, and which was confined and surgically resected (or treated with other mo-dalities) with curative intent and unlikely to im-pact survival during the duration of the study.
13. Participant is pregnant or lactating
14. Participants who have had prior allogeneic stem cell transplant.
15. Participants with symptomatic amyloidosis, ac-tive POEMS syndrome (polyneuropathy, or-ganomegaly, endocrinopathy, monoclonal plasmaproliferative disorder, skin changes) or active plasma cell leukaemia at the time of screening.
16. Participants with any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including lab abnormalities) that could interfere with participant's safety, ob-taining informed consent or compliance to the study procedures.
17. Subject is known to be seropositive for human immunodeficiency virus (HIV) or hepatitis B (defined by a positive test for hepatitis B sur-face antigen (HBsAg) or antibodies to hepatitis B surface and core antigen (anti HBs and anti HBc respectively), or hepatitis C (anti-HCV an-tibody positive or HCV RNA quantitation posi-tive).
18. Current immune or inflammatory conditions re-quiring immunosuppressive treatment (e.g. systemic lupus erythematosus, rheumatoid ar-thritis).
19. Subject must not have received any live vac-cines within 8 weeks prior to first dose of study treatment.
20. Subject must not use or anticipate the use of prohibited medications or foods during study participation.
21. Subject does not have a history of or show any signs of known meningeal/central nervous sys-tem involvement by myeloma.
22. Evidence of other clinically significant uncon-trolled condition(s) that is likely to interfere with the study proce-dures or results, or that in the opinion of the investigator, would constitute a hazard for the participation in this study.
23. Subject is known or suspected of not being able to comply with the study protocol. Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being) or that could prevent, limit or confound the pro-tocol-specified assessments.
24. Treatment with any of the following within 7 days prior to the first dose of study drug:

    1. moderate or strong cytochrome P450 3A (CYP3A) inhibitors
    2. moderate or strong CYP3A inducers
25. Administration or consumption of any of the fol-lowing within 3 days prior to the first dose of study drug:

    1. grapefruit or grapefruit products
    2. Seville oranges (including marmalade con-taining Seville oranges)
    3. star fruit
26. Participation in any other clinical trial (with the exclusion of observational studies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II dose (RP2D) | approx. 9 months
  Establishment of Recommended Phase II dose (RP2D), Evaluation of safety profile, including maximum tolerated dose

SECONDARY OUTCOMES:
Overall Response Rate | through study completion, an average of 2 years
  Overall Response Rate
Minimal residual disease (MRD) negativity | through study completion, an average of 2 years
  Minimal residual disease (MRD) negativity rate and duration
Progression free survival (PFS) | through study completion, an average of 2 years
  Progression free survival (PFS)
Duration of response (DOR) | through study completion, an average of 2 years
  Duration of response (DOR)

CONTACTS AND LOCATIONS:
Overall Officials: Katja Weisel, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (5):
- Germany (5):
  - University Medical Center Hamburg-Eppendorf, Hamburg, Ham
  - Klinikum Chemnitz, Chemnitz
  - Uniklinik Heidelberg, Heidelberg
  - UKSH Lübeck, Lübeck
  - Uniklinkum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No